CLINICAL TRIAL: NCT00370760
Title: Oral Colchicine Combined With Intravitreal Infusion of Dexamethasone, LMW Heparin and 5-FU for Management of Proliferative Vitreoretinopathy (PVR)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8404
Record Dates: First submitted 2006-08-30; First posted 2006-09-01 (Estimated); Last update posted 2008-06-26 (Estimated); Status verified 2008-06

CONDITIONS: Proliferative Vitreoretinopathy
Keywords: PVR; Oral colchicine; Dexamethasone; low molecular weight heparin; 5-FU
MeSH Terms: conditions — Vitreoretinopathy, Proliferative | interventions — Colchicine; Dexamethasone; Heparin, Low-Molecular-Weight; Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: oral colchicine, dexamethasone, low molecular weight heparin, 5-FU
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: oral colchicine, dexamethasone, low molecular weight heparin, 5-FU
  Arms: 1
Drug: placebo
  Arms: 2

SUMMARY:
To evaluate the efficacy of oral colchicine combined with intraoperative infusion of dexamethasone, low molecular weight heparin and 5-FU during vitrectomy for management of established proliferative vitreoretinopathy (PVR)

ELIGIBILITY:
Inclusion Criteria:

* Cases with rhegmatogenous retinal detachment complicated by PVR grade C

Exclusion Criteria:

* History of pars plana vitrectomy for PVR grade C
* History of silicone oil injection
* History of ocular trauma
* Diabetic retinopathy
* Glaucoma
* Giant retinal tear

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2006-09

PRIMARY OUTCOMES:
Retinal reattachment rate

SECONDARY OUTCOMES:
PVR recurrence,
macular pucker,
reoperation,
ocular hypotony,
visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ahmadieh, MD, Principal Investigator — Ophthalmic Research Center of Shaheed Beheshti Medical University
Locations (1):
- Hamid Ahmadieh, MD, Tehran, Tehran Province, Iran